CLINICAL TRIAL: NCT00599235
Title: Effects of the Selective Phosphodiesterase Type 5 Inhibitor Sildenafil Citrate on Exercise Capacity and Vascular Function in Hypertensive Subjects
Brief Title: Sildenafil and Exercise Capacity in Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Marise Bucukoglu, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: LREC/2004/4/13; LREC/2004/4/13
Record Dates: First submitted 2008-01-07; First posted 2008-01-23 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2008-01

CONDITIONS: Hypertension
Keywords: Hypertension; Exercise capacity; PDE5 inhibitors
MeSH Terms: conditions — Hypertension | interventions — Sildenafil Citrate; Hydralazine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: sildenafil; Drug: hydralazine; Drug: placebo
- 2 (Active Comparator)
  Interventions: Drug: sildenafil; Drug: hydralazine; Drug: placebo

INTERVENTIONS:
Drug: sildenafil — 50mg 3 times daily for 7 days
  Other Names: Viagra
Drug: hydralazine — 25mg 3 times daily for 7 days
Drug: placebo — 3 times daily for 7 days

SUMMARY:
Hypertension (persistently elevated blood pressure) is a major risk factor for heart disease and stroke. Hypertensive individuals show a reduced exercise capacity, which is present from a very early stage and contributes to their increased cardiovascular risk. Sildenafil belongs to a class of drugs called phosphodiesterase type 5 (PDE5) inhibitors, and it works by enhancing the effects of nitric oxide, a substance that dilates blood vessels and increases blood flow. We hypothesize that sildenafil, because of its effect on nitric oxide and blood flow, will improve exercise capacity in hypertensive patients. Therefore, the main aim of the study is to investigate the effects of PDE5 inhibition on exercise capacity and vascular function in hypertension, and to compare these effects in hypertensive patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Male (age range: 18 - 70 years)
* Appropriate blood pressure range
* Hypertensive - Systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg
* Controls - Systolic BP <140 mmHg and diastolic BP <90mmHg
* Written informed consent

Exclusion Criteria:

* Female
* History of coronary artery, cerebrovascular or peripheral vascular disease within the last 6 months
* Total cholesterol >6.5 mmol/L
* Current alcohol abuse
* Diabetes mellitus
* Asthma
* Taking any anti-hypertensive, vasoactive or endothelial function modifying drugs which cannot be withdrawn for the purpose of the study
* ECG evidence of clinically significant arrhythmia or cardiac ischaemia
* Clinically significant abnormality on screening blood test
* Contraindication to strenuous exercise
* Current involvement in other research projects
* Other clinically relevant conditions
* Lack of written informed consent

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2) during exercise | 1 week of treatment

SECONDARY OUTCOMES:
Exercise systolic blood pressure | Maximal exercise
Pulse wave velocity and pulse wave analysis | Before and after maximal exercise

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M Attinà, MD, Principal Investigator — University of Edinburgh; David J Webb, MD, Study Director — University of Edinburgh
Locations (1):
- University of Edinburgh - Western General Hospital, Edinburgh, United Kingdom